CLINICAL TRIAL: NCT04832399
Title: Tysabri in Early Relapsing Remitting Multiple Sclerosis Patients - TYPIFI (Tysabri Patient Initiation After Failure of the Initial DMT)
Brief Title: Study of Tysabri in Early Relapsing Remitting Multiple Sclerosis Participants
Acronym: TYPIFI
Status: Completed | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: PRT-TYS-12-10409
Record Dates: First submitted 2021-03-16; First posted 2021-04-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Relapsing Remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Natalizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Natalizumab: Natalizumab 300 mg is administered by intravenous infusion once every 4 weeks.
  Interventions: Drug: Natalizumab

INTERVENTIONS:
Drug: Natalizumab — As described in the treatment arm.
  Other Names: Tysabri; BG00002

SUMMARY:
The purpose of this study is to evaluate the impact of an early treatment with Natalizumab on the management of the progressive nature of Relapsing Remitting Multiple Sclerosis (RRMS).

ELIGIBILITY:
Key Inclusion Criteria:

* Documented diagnosis of Relapsing Remitting Multiple Sclerosis (McDonald 2010 Criteria).
* EDSS ≤ 3.0.
* Must fulfill Tysabri indication (relapse and MRI criteria).
* Decision to start treatment with Natalizumab must precede enrollment.
* Up to four natalizumab infusions.

Key Exclusion Criteria:

* Any prior treatment with Natalizumab.
* Prior imunossupressive treatment (Mitoxantrone, Azathioprine, Methotrexate, Cyclophosphamide, Mycophenolate, Cladribine, Rituximab).
* Contraindications to treatment with Natalizumab.
* History of Progressive Multifocal Leukoencephalopathy (PML) or other opportunistic infections, or an increased risk for such infections.
* Immunocompromised at the time of enrollment. Known active malignancies.
* Inability to comply with study requirements.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Participants diagnosed with relapsing remitting multiple sclerosis (RRMS) that have been prescribed natalizumab under standard clinical care.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2013-11-12 (Actual); Primary Completion 2023-10-02 (Actual); Study Completion 2023-10-02 (Actual)

PRIMARY OUTCOMES:
Overall Disease-Free Status at Month 12 | Month 12
Clinical Disease-Free Status at Month 12 in Comparison to the Previous Year | Month 12
Annualized Relapse Rate at Month 12 in Comparison to the Previous Year | Month 12

SECONDARY OUTCOMES:
Overall Disease-Free Status at Months 24, 36 and 48 | Months 24, 36 and 48
Clinical Disease-free Status Every 6 Months | Every 6 months (Up to 48 months)
Annualized Relapse Rate (ARR) | Months 12, 24, 36 and 48
Change From Baseline in Sustained Expanded Disability Status Scale (EDSS) Score (24-week Sustained) | Months 12, 24, 36 and 48
  The EDSS is used to quantify disability due to symptoms of MS and to track changes in disability status over time. Scores range from 0 (normal neurological exam) to 10 (death due to multiple sclerosis).
MRI measures: T2, T1, T1 with Gadolinium (Gd) | Months 12, 24, 36 and 48
Cognitive Impairment Using Symbol Digit Modalities Test (SDMT) | Months 12, 24, 36 and 48
Change From Baseline in Ability to Work and Productivity as Assessed by Work Productivity and Activity Impairment (WPAI) Questionnaire | Months 12, 24, 36 and 48
  The WPAI questionnaire is a validated instrument to measure impairments in work and activities. The WPAI yields four types of scores: 1. Absenteeism (work time missed) 2. Presenteesism (impairment at work / reduced on-the-job effectiveness) 3. Work productivity loss (overall work impairment / absenteeism plus presenteeism) 4. Activity Impairment. WPAI outcomes are expressed as impairment percentages ranging from 0-100%, with higher numbers indicating greater impairment and less productivity.
Quality of life (QoL) Assessed Using Fatigue Severity Scale | Months 12, 24, 36 and 48
  The FSS is a self-assessment questionnaire that provides a score as a measurement of the severity of fatigue. It consists of 9 questions scored from 1 to 7. A low value (e.g., 1); indicates strong disagreement with the statement, whereas a high value (e.g., 7); indicates strong agreement. A total score of 36 or more suggests presence of fatigue.
QoL assessed using Multiple Sclerosis Functional Composite (MSFC) Test | Months 12, 24, 36 and 48
  MSFC has 2 component- timed 25-foot walk (T25FW) and 9-hole peg test (9HPT) [dominant and nondominant hands]. The MSFC Z-score is calculated by creating Z-scores for each component of the MSFC and averaging them to create an overall composite score. MSFC Z-score = (Z25-foot-walk + Z9HPT-2)/2, where Zj refers to Z-scores of component j. A Z-score represented the number of standard deviations participant's test result was higher (Z >0) or lower (Z <0) than the average test result (Z = 0) from the reference population. Higher scores indicate better outcomes.
QoL Assessed Using Beck Depression Inventory, 2nd Edition (BDI-II) | Months 12, 24, 36 and 48
  BDI-II Scale is a 21-item self-reported questionnaire which measures the existence and severity of symptoms of depression. Each of the 21 items on BDI-II tool represents a depressive symptom. The symptoms are each scored on a 4-point Likert scale of 0 to 3 (0=symptom is absent; 3=symptom is severe). Scores for each symptom are added up to obtain the total scores for all 21 items. Total score ranges from 0-63; of which 0-8 is considered no depression, 0-13 is minimal depression, 14-19 is mild depression, 20-28 is moderate depression and 29-63 is severe depression.
QoL Assessed Using Multiple Sclerosis Impact Scale (MSIS-29) | Months 12, 24, 36 and 48
  MSIS-29 is a brief self-administered instrument measuring physical (20 items) and psychological (9 items) impact of Multiple Sclerosis (MS). Each of the 29 items on MSIS-29 tool is a question that ask for participants views about the impact of MS on their day to day lives. Each item is scored on 1 to 5 (1=Not at all; 5=Extremely).

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (18):
- Portugal (18):
  - Research Site, Amadora
  - Research Site, Angra do Heroísmo
  - Research Site, Aveiro
  - Research Site, Braga
  - Research Site, Coimbra
  - Research Site, Faro
  - Research Site, Funchal
  - Research Site, Guimarães
  - Research Site, Leiria
  - Research Site, Lisbon
  - Research Site, Loures
  - Research Site, Matosinhos Municipality
  - Research Site, Penafiel
  - Research Site, Porto
  - Research Site, Santa Maria da Feira
  - Research Site, Setúbal
  - Research Site, Viana do Castelo
  - Research Site, Vila Nova de Gaia